CLINICAL TRIAL: NCT04460105
Title: A Phase 1b, Randomized, Double-blind, Single and Repeat Dosing Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Lanadelumab When Added to Standard-of-Care in Subjects Hospitalized With COVID-19 Pneumonia
Brief Title: Lanadelumab in Participants Hospitalized With COVID-19 Pneumonia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was withdrawn due to challenges in site recruitment and lack of patient enrollment
Sponsor: Shire (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TAK-743-1002
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — lanadelumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lanadelumab (Experimental): Participants receive 300 milligram (mg) of lanadelumab intravenous (IV) infusion on Day 1 during Cohort 1 (single dose cohort) and on Day 1 and Day 4 during Cohort 2 (repeat-dose cohort).
  Interventions: Drug: Lanadelumab
- Placebo (Placebo Comparator): Participants will receive placebo matching IV infusion on Day 1 during Cohort 1 (single dose cohort) and on Day 1 and Day 4 during Cohort 2 (repeat-dose cohort).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lanadelumab — Participants will receive 300 mg of lanadelumab IV infusion on Day 1 and Day 4.
  Other Names: SHP643; TAK-743; DX-2930
  Arms: Lanadelumab
Other: Placebo — Participants will receive placebo matching IV infusion on Day 1 and Day 4.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetic and pharmacodynamics of lanadelumab administered by intravenous (IV) infusion when added to standard-of-care (SoC) in adults hospitalized with COVID-19 pneumonia.

DETAILED DESCRIPTION:
This study consists of two cohorts (Cohort 1 [Single-dose Cohort], and Cohort 2 [Repeat-dose Cohort]). Up to approximately 24 participants will be enrolled in this study, in which up to 12 participants may be enrolled into Cohort 1. However, Cohort 1 will be closed upon implementation of Amendment 2. Approximately 12 participants will be enrolled in Cohort 2. Participants will be randomized in 3:1 ratio (9 lanadelumab: 3 placebo) in each Cohort.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years of age or older at the time of signing of the informed consent form (ICF).
* Hospitalized with evidence of COVID-19 pneumonia defined as:

  1. Severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) infection documented with polymerase chain reaction (PCR) of any specimen; e.g. respiratory, blood, urine, stool, other body fluid
  2. Presence of respiratory distress as indicated by peripheral capillary oxygen saturation (SpO2) lesser than or equal to (=<) 93 percent (%) on room air or respiratory rate greater than or equal to (>=) 30 breaths per minute (breaths/min).
* The participant (or a legally acceptable representative) has provided written informed consent approved by the institutional review board (IRB)/ independent ethics committee (IEC) before any study-specific procedures are performed.
* Agree to adhere to the protocol-defined schedule of treatments, assessments, and procedures.

Exclusion Criteria:

* Invasive mechanical ventilation (IMV) extracorporeal membrane oxygenation (ECMO) or with evidence of severe respiratory distress such that IMV/ECMO is imminent within 12 hours of randomization.
* Where, in the opinion of the investigator, progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatments.
* Requiring vasopressor support (use of fluid support is not exclusionary)
* Known or suspected venous thromboembolism.
* Known or suspected hypersensitivity to lanadelumab or any of its excipients.
* Dosing with an investigational drug or exposure to an investigational device within 4 weeks prior to screening.
* Previous (within 3 months of screening) or current use of immunomodulators (e.g. methotrexate, azathioprine, 6-mercaptopurine, tumor necrosis factor [TNF] alpha inhibitor, Janus kinase [JAK] inhibitor, alpha-integrin).
* Previous (within 3 months of screening) or current use of plasma kallikrein inhibitor or bradykinin receptor blocker.
* Use of supplemental oxygen for a medical condition prior to receiving COVID-19 diagnosis.
* Previously diagnosed with acquired immunodeficiency syndrome (AIDS).
* Active tuberculosis or clinical suspicion of latent tuberculosis.
* Any of the following laboratory abnormalities at screening:

  1. Hemoglobin <= 8 grams per deciliter (g/dL)
  2. White blood cells <= 3000/ microliters (μL)
  3. Platelets <= 75,000/μL
  4. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >= 3×upper limit of normal (ULN); alkaline phosphatase (ALP) >= 3×ULN; or total bilirubin greater than (>) 2×ULN (unless the bilirubin elevation is a result of Gilbert's syndrome)
  5. Creatinine >= 2×ULN
* Pregnant or breastfeeding.
* Any significant condition (any surgical or medical condition) that, in the opinion of the investigator or sponsor, may compromise their safety or compliance, preclude the successful conduct of the study, or interfere with interpretation of the results (e.g. significant pre-existing illness or other major comorbidities that the investigator considers may confound the interpretation of study results).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-31 (Estimated); Primary Completion 2021-01-27 (Estimated); Study Completion 2021-01-27 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment emergent adverse events (TEAEs) | From start of study drug administration to follow-up (up to Day 29)
  Treatment-emergent adverse events are defined as Adverse events (AEs) with onset at the time of or following the start of treatment with study medication, or medical conditions present prior to the start of treatment but increasing in severity or relationship at the time of or following the start of treatment. SAE is any untoward clinical manifestation of signs, symptoms or outcomes (whether considered related to investigational product or not and at any dose: results in death, is lifethreatening, requires inpatient hospitalization or prolongation of hospitalization, results in persistent or significant disability/incapacity, congenital abnormality/birth defect, an important medical event. AESI will include hypersensitivity reactions, events of disordered coagulation such as bleeding AESI, hypercoagulable AESI. Number of participants with TEAEs including AESI and SAE will be assessed.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Plasma Concentrations of Lanadelumab | Single-dose Cohort: Pre-dose, 1, 24, 72, 144, 216, 336 hours post-dose; Repeat-dose Cohort: Pre-dose, 1, 24, 72, 73, 144, 216, 336 hours post-dose
  Pharmacokinetic plasma concentrations of lanadelumab after a single and repeat intravenous (IV) doses will be assessed.
Percentage Change from Baseline in Plasma Kallikrein Activity (pKal) | Single-dose Cohort: Pre-dose, 1, 24, 72, 144, 216, 336 hours post-dose; Repeat-dose Cohort: Pre-dose, 72, 144, 216, 336 hours post-dose
  Percentage change from baseline in pKal activity to assess pharmacodynamics (PD) of lanadelumab.
Percentage Change from Baseline in Cleaved High Molecular Weight Kininogen (cHMWK) | Single-dose Cohort: Pre-dose, 1, 24, 72, 144, 216, 336 hours post-dose; Repeat-dose Cohort: Pre-dose, 72, 144, 216, 336 hours post-dose
  Percentage change from baseline in cHMWK levels to assess PD of lanadelumab.
Percentage Change from Baseline in Functional C1-Inhibitor (C1-INH) | Single-dose Cohort: Pre-dose, 1, 24, 72, 144, 216, 336 hours post-dose; Repeat-dose Cohort: Pre-dose, 72, 144, 216, 336 hours post-dose
  Percentage change from baseline in functional C1-INH levels to assess PD of lanadelumab.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda Development Center Americas, Inc.

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/